CLINICAL TRIAL: NCT05214937
Title: A Distance-based, Randomized Controlled Trial for Reducing Sedentary Behaviour Among Prostate Cancer Survivors
Brief Title: A Intervention for Reducing Sedentary Behaviour Among Prostate Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Linda Trinh, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 28981
Record Dates: First submitted 2021-12-15; First posted 2022-01-31 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Sedentary Behavior; Cancer of Prostate
Keywords: distance-based; sedentary behavior; physical activity; cancer survivorship
MeSH Terms: conditions — Sedentary Behavior; Prostatic Neoplasms; Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomization will be performed using a stratified randomization scheme via REDCap. The sequence will be random permutated blocks of varying sizes, stratified by ADT use (ADT vs. no ADT). PCS will be assigned in a 1:1 ratio to one of two groups. Randomization codes will be kept in a pre-made digital file that is separate from other study records.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is not possible to blind participants to their group allocation. Coordinating RAs will be the primary individuals responsible for scheduling all data collection assessments.
  They will attempt to book all 3 assessments with same research assistant outcome assessor who meets the following criteria:
  * Are not a movement specialist delivering one-on-one behavioural counselling
  * Are not a movement specialist delivering a group webinar
  * Are not aware of participant's group allocation
  Any cases of unblinding will be noted in a Protocol Deviation Log.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be provided with a FitBit Inspire 2 and assigned a movement specialist. They will be asked to monitor their daily steps over the 12-week intervention period. Participants will attend 6 remotely-delivered behaviour change sessions (4 one-on-one sessions with their movement specialist, 2 group-based webinars). Sessions will be delivered bi-weekly and last ~30 minutes.
  Interventions: Behavioral: Intervention
- Fitbit Only (Active Comparator): Participants will be provided with a FitBit Inspire 2 and access to publicly available resources about active living (e.g., 24-hour movement guidelines).
  Interventions: Behavioral: FitBit Only

INTERVENTIONS:
Behavioral: Intervention — During the first two weeks (baseline), participants will be asked to maintain their regular movement routine to set a baseline daily average step count. Phases I-III will involve self-regulatory strategies (e.g., action planning), address reducing/interrupting sedentary time, and step counts. Participants will be encouraged to increase their steps by 1000 steps/day from the baseline phase during each subsequent phase (i.e., 3000 steps above baseline by Phase III). Phases IV-V will be a maintenance phase through which participants will be encouraged to maintain 3000 steps per day above baseline. The sessions will be grounded within the Multi-Process Action Control Framework and address perceived capability/opportunity and instrumental/affective attitudes. The 1-on-1 sessions will focus on regulation (action & coping planning, social support, goal setting) and reflexive processing (self-regulation, habit). The final one on one session will be a booster session to revisit previous topics.
  Arms: Intervention
Behavioral: FitBit Only — Participants will be provided with a FitBit Inspire 2 and access to publicly available resources about active living. They will receive a FitBit orientation session with a movement specialist prior to the 12-week control period.
  Arms: Fitbit Only

SUMMARY:
This randomized controlled trial (RCT) will aim to examine the effect of a 12-week behavioural intervention on changing the sedentary behaviours (SB) of prostate cancer survivors (PCS) compared to a control group (FitBit-only group). PCS in the intervention group will receive a FitBit and 6 behavioural support sessions with a movement specialist guided by behavioural theory (i.e., the Multi-Process Action Control [M-PAC]). The FitBit-only group will only receive a FitBit and access to public health resources on physical activity (PA). The primary purpose of this study is to determine the efficacy of the intervention on changing SB of PCS immediately following the 12-week intervention and 6-months later. It is hypothesized that that the intervention will decrease their SB compared to the FitBit-only control condition at both timepoints. This trial will also examine the effect of the intervention on changing PA, motivational outcomes from the M-PAC framework, sleep quality, social support, physical function, quality of life, fatigue, disability and mental health compared to the active control condition.

DETAILED DESCRIPTION:
Many prostate cancer survivors (PCS) suffer from long-term side effects well beyond treatment, such as urinary incontinence, erectile dysfunction, fatigue, depression, and anxiety. Supportive care interventions are needed to reduce the chronic effects of cancer and its treatment during the transition into survivorship. Physical activity (PA) has a positive impact on many clinical outcomes, including improved quality of life (QoL), cancer-specific mortality, and reducing treatment-related toxicities among PCS. Despite this, few PCS achieve current PA guidelines and there is a significant decrease in PA during and following treatment. PCS spend most of their day sedentary (i.e., 69% of waking hours) or engaged in light-intensity PA (LPA; 30% of waking hours), therefore focusing on reducing sedentary behaviour (SB) among PCS may be a more feasible intervention approach than supervised exercise. SB is defined as any waking behaviour characterized by a low energy expenditure (i.e., ≤1.5 resting metabolic equivalents) while in a sitting, reclining, or lying down posture. Despite the growing evidence that reducing SB can result in better health outcomes for cancer survivors, there are no known effective strategies aimed at reducing SB and replacing it with PA among PCS.

It is important that behavioural interventions are informed by theory, as theory-driven approaches are crucial for facilitating the adoption and maintenance of behaviour change. The Multi-Process Action Control (M-PAC) framework, a theoretical framework developed from PA behaviour change research specifically, suggests a layered, progressive approach to behaviour change where an individual moves from intention formation to adoption of action control and onto maintenance of action control. Intention formation is predicated on initiating reflective processes (i.e., instrumental attitude and perceived capability). Reflective processes are hypothesized to influence intention formation and initiate regulatory processes to enact this intention (i.e., affective attitude and perceived opportunity). The translation of intention into PA (i.e., action control) is determined partially by regulatory processes (e.g., action planning, coping planning, self-monitoring, social support) during the initial adoption of the behaviour. Continuation of PA action control is thought to include the addition of reflexive processes (e.g., habit) for long-term PA maintenance. This is a useful approach for PA and SB behaviour change interventions as it highlights processes for several stages of change including adoption and maintenance.

Previously supervised interventions have demonstrated success in increasing PA behaviours among cancer survivors but, distance-based interventions make an attractive alternative as they have extended reach due to potentially easier access and lower cost. Wearable activity monitors (e.g., FitBit) have been a successful SB and PA self-management intervention tool for cancer survivors. A previous pilot study conducted by our research group examined the feasibility of an unguided mhealth application (RiseTx) for reducing SB and increasing MVPA among PCS undergoing androgen deprivation therapy (ADT). PCS were given an activity tracker, access to the RiseTx mhealth web application which deployed a range of behaviour change support tools to reduce SB, and a goal of increasing step counts by 3,000 daily steps above baseline levels over 12-weeks. The RiseTx mhealth application was successful in reducing device-measured SB by 455 minutes/week and increasing MVPA by 44 minutes/week, as well as increasing steps by 1535 between baseline and post-intervention. Building upon this successful pilot study, the current RCT will harness the many lessons learned during the implementation of the RiseTx mhealth application. As an extension of this prior work, this updated iSTRIDE intervention will provide additional synchronous behavioural support aligned with processes in the M-PAC framework through videoconferencing, to reduce SB.

The multi-site, two-arm RCT will test the efficacy of this updated intervention on changing SB and PA in PCS. The primary objective is to determine the effects of the 12-week intervention (i.e., FitBit + behavioural counselling) compared to a control condition (FitBit + public resources) in reducing sitting time in PCS. It is hypothesized that that the intervention group will decrease their SB compared to the FitBit-only control condition at post-intervention (12 weeks) and 6-month follow-up. Secondary objectives of this trial are to determine the effects of the intervention on secondary outcomes including changes in MVPA, LPA, motivational outcomes from the M-PAC framework, sleep quality, social support, physical function and patient reported outcomes (i.e., QoL, fatigue, disability and mental health) compared to the FitBit-only control condition.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Diagnosed with localized or asymptomatic metastatic primary prostate cancer
* Not currently undergoing radiation or chemotherapy
* Proficient in English
* Not physically active (self report <150 minutes of moderate-to-vigorous physical activity per week)
* Self-report >8 hours of daily sedentary behaviour
* In the contemplation or preparation stage for motivational readiness to change as determined by the Stages of Change Questionnaire
* Access to a smartphone, tablet, or computer
* No cardiac contraindications (e.g., unstable angina, arrhythmia, heart failure, aortic stenosis)
* Medical clearance from a primary health care provider (if necessary)
* Currently residing in Canada

Exclusion Criteria:

* Not planning to live in Canada for the next 12 months
* A medical condition that prohibits walking (e.g., severe knee or hip arthritis)
* Presence of other primary or recurrent invasive cancer (i.e., other than non-melanoma skin cancer)
* Have had a prior fall within the last 12-months
* Use a gait aid device

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in sedentary behaviour as assessed by activPAL inclinometers | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Objectively-assessed sedentary behaviour will be assessed with activPAL inclinometers. The activPALs will be waterproofed and participants will be asked to wear the device in the mid-line of their right thigh for 7 days (24 hours per day). Participants will complete a wear log to identify sleep and non-wear periods. Total daily minutes of sedentary behaviour will be collected from the devices.

SECONDARY OUTCOMES:
Change in Self-reported Sedentary Behaviour as assessed by the Longitudinal Aging Study Amsterdam | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Self-reported sedentary behaviour will be assessed with the Longitudinal Aging Study Amsterdam (LASA) sedentary behaviour questionnaire. It assesses weekday and weekend sedentary time across 10 domains. The time (hours/minutes) in each domain is summed to determine a total amount of sedentary time.
Change in Self-Reported Physical Activity assessed by the Godin Leisure Time Exercise Questionnaire | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Self-reported leisure time exercise will be assessed using the Godin Leisure Time Exercise Questionnaire. Participants will self-report the frequency and duration of light, moderate, and vigorous leisure-time exercise. This will be used to calculate a total leisure activity score (higher score indicates higher volumes of activity). The GLTEQ is a valid and reliable measure of exercise among oncology populations.
Change in Objectively-assessed Physical Activity as assessed by activPAL inclinometers | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Objectively-assessed activity will be assessed with the activPALs. Minutes of activity at a cadence >100 steps per minute will be considered moderate-to-vigorous physical activity.

OTHER OUTCOMES:
Change in Reflective Motivational Processes | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Perceived capability and opportunity will be assessed using a modified version of the Rhodes et al., (2006) measures of ability and opportunity. These constructs are measured through six statements (3 addressing ability and 3 addressing opportunity) regarding confidence and control over engaging in light physical activity to replace sedentary behaviour and scored using a 5-point likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Possible scores range from a 3-15 points with higher scores indicating more favorable perceptions of opportunity and ability.
  Instrumental attitudes and affective judgements will be assessed using a modified version of the Rhodes and Courneya (2003) instrumental and affective attitude measure using a 7-point Likert scale (extremely disagree to extremely agree).
Change in Regulatory Motivational Processes | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Regulatory processes will be measured through decisional intentions and behavioural regulation (i.e.,planning and monitoring). Decisional intentions will be measured using the following questions "I intend to engage in regular light physical activity _ times per week during the next 12 weeks", "I intend to break up my sitting time _ times per weekday during the next 12 weeks." and "I intend to break up my sitting time ________ times per weekend day during the next 12 weeks."
  Behavioural regulation was measured using a modified version of the Sniehotta et al., (2005) planning questionnaire which assesses goal setting, action and coping planning, self-monitoring and scheduling on a 6-item scale. Each item is scored on a 5-point likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 6-30 points with higher scores indicating better self-regulation.
Change in Reflexive Motivational Processes | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Reflexive processes will be measured through habit formation with the Self-Report Behavioural Automaticity Index from Gardner et al., (2012). Items are scored on a 5-point likert scale (1-strongly disagree to 5-strongly agree) summed to create a total score. Total scores can range from 4-20 points where higher scores indicate a behaviour is more habitual.
Change in Disease-Specific Quality of Life as assessed by the Functional Assessment of Cancer Therapy | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Disease-specific quality of life will be assessed with the reliable and well-validated Functional Assessment of Cancer Therapy (FACT)-General which consists of physical well-being (PWB), functional well-being (FWB), emotional well-being (EWB), and social well-being (SWB) subscales. The FACT-Fatigue (FACT-Fatigue) scale includes the 27 items from the FACT-General scale plus the 13-item fatigue subscale. On all scales, higher scores indicate better QoL and less symptoms. Scores range from 0-108 and 0-156 for the FACT-General and FACT-Fatigue, respectively. Lower scores indicate a better quality of life.
Change in Health-related Quality of Life as assessed by the Short Form-12 | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  General health-related quality of life will be measured using the Short Form-12 (SF-12). The SF-12 is a 12-item, shortened version of the SF-36 assessing physical functioning, bodily pain, role functioning, emotional well-being, social functioning, energy/fatigue, and health perceptions. It also includes a single item that provides an indication of perceived change in health. The SF-12 has good test-retest reliability correlations of 0.89 and 0.76 for the physical and mental component score, respectively. Additionally, scores from the SF-12 is highly correlated with scores from the complete SF-36 questionnaire. Higher scores indicate better quality of life. The SF-12 has been previously used in cancer populations.
Change in Mental Health as assessed by the Hospital Anxiety and Depression Scale | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Mental health, including anxiety and depression, will be assessed with the Hospital Anxiety and Depression Scale (HADS). The HADS is a 14-item instrument comprised of an anxiety subscale score (HADS-A), a depression subscale score (HADS-D) and a total score (HADS-T), where higher scores indicate higher distress. Each item on the HADS is rated on a 4-point Likert scale, where 0 = 'not at all' and 3 = 'yes, definitely.'
Internet & Technology Use as assessed by the eHEALS eHealth literacy scale | Baseline
  Technology literacy (measured at baseline only) will be assessed using a modified version of the 8-item eHEALS ehealth literacy scale. The eHEALS measures combined knowledge, comfort, and perceived skills at finding, evaluating, and applying electronic health information to health problems. It will be adapted to assess confidence in using and finding online information related to sedentary time and physical activity. Items will be rated using a 5-point Likert scale (strongly disagree-strongly agree). Scores range from 8-40 which higher scores representing greater self-perceived eHealth literacy.
  10 researcher-generated questions will assess general patterns of internet and social media use, including methods used to access the internet and social media, frequency of use, devices owned and types of social media accounts owned, as well as use of internet and social media for information related to sedentary time and physical activity.
Change in Health & Disability as assessed by the WHODAS 2.0 | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Disability will be assessed using the self-administered 12-item World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0). This questionnaire is used to assess functioning in six major life domains (e.g., cognition, mobility, self-care, getting along, life activities, and participation). Simple scoring method will be used to sum the 12 items to create a Global Disability total score that will be used to describe the functional limitation of prostate cancer survivors. The scores for each item ranges from 1 (none) to 5 (extreme). Scores range from 1 to 60, higher scores represent greater disability.
Program Feedback | Post-Intervention (12-weeks)
  A participant satisfaction survey will be administered post 12-week intervention to assess the acceptability of the intervention using research generated, closed response questions that ask: "Did the movement specialist effectively demonstrate constructive feedback throughout the Program"; "Was the workbook information and easy to follow?". The survey will assess the burden of the program and feedback about the manual, counselling sessions, and overall study experience. Likert scales ranging from 1 (not at all) to 7 (very much) will be used.
Physical Function as assessed by the 30 second sit to stand | Baseline, Post-Intervention (12-weeks), 6-month Follow Up
  Lower body strength will be assessed with the 30-second sit to stand test. Participants will set up an armless chair against a wall or stable surface within view of the camera. Participants will start with their arms crossed over their chest, in the middle of the chair with their back straight, and feet flat on the floor. The participant will be instructed to stand fully then return to the start position as many times as they can in the 30-second assessment window. Study staff will oversee timing and counting the number of repetitions. Repetitions will only be scored if the participant touches the chair at the bottom of the movement and stand up completely straight at the top of the movement. Higher scores represent greater physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Trinh, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amireault S, Godin G, Lacombe J, Sabiston CM. The use of the Godin-Shephard Leisure-Time Physical Activity Questionnaire in oncology research: a systematic review. BMC Med Res Methodol. 2015 Aug 12;15:60. doi: 10.1186/s12874-015-0045-7. PMID 26264621
- [Background] Andrews G, Kemp A, Sunderland M, Von Korff M, Ustun TB. Normative data for the 12 item WHO Disability Assessment Schedule 2.0. PLoS One. 2009 Dec 17;4(12):e8343. doi: 10.1371/journal.pone.0008343. PMID 20020047
- [Background] Brucker PS, Yost K, Cashy J, Webster K, Cella D. General population and cancer patient norms for the Functional Assessment of Cancer Therapy-General (FACT-G). Eval Health Prof. 2005 Jun;28(2):192-211. doi: 10.1177/0163278705275341. PMID 15851773
- [Background] Burrell AMG, Allan JL, Williams DM, Johnston M. What do self-efficacy items measure? Examining the discriminant content validity of self-efficacy items. Br J Health Psychol. 2018 Sep;23(3):597-611. doi: 10.1111/bjhp.12306. Epub 2018 Mar 8. PMID 29520897
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Djukanovic I, Carlsson J, Arestedt K. Is the Hospital Anxiety and Depression Scale (HADS) a valid measure in a general population 65-80 years old? A psychometric evaluation study. Health Qual Life Outcomes. 2017 Oct 4;15(1):193. doi: 10.1186/s12955-017-0759-9. PMID 28978356
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Gardner B, Abraham C, Lally P, de Bruijn GJ. Towards parsimony in habit measurement: testing the convergent and predictive validity of an automaticity subscale of the Self-Report Habit Index. Int J Behav Nutr Phys Act. 2012 Aug 30;9:102. doi: 10.1186/1479-5868-9-102. PMID 22935297
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Kozey-Keadle S, Libertine A, Lyden K, Staudenmayer J, Freedson PS. Validation of wearable monitors for assessing sedentary behavior. Med Sci Sports Exerc. 2011 Aug;43(8):1561-7. doi: 10.1249/MSS.0b013e31820ce174. PMID 21233777
- [Background] Lyden K, Keadle SK, Staudenmayer J, Freedson PS. The activPALTM Accurately Classifies Activity Intensity Categories in Healthy Adults. Med Sci Sports Exerc. 2017 May;49(5):1022-1028. doi: 10.1249/MSS.0000000000001177. PMID 28410327
- [Background] Lynch BM, Dunstan DW, Winkler E, Healy GN, Eakin E, Owen N. Objectively assessed physical activity, sedentary time and waist circumference among prostate cancer survivors: findings from the National Health and Nutrition Examination Survey (2003-2006). Eur J Cancer Care (Engl). 2011 Jul;20(4):514-9. doi: 10.1111/j.1365-2354.2010.01205.x. Epub 2010 Jun 29. PMID 20597954
- [Background] Norman CD, Skinner HA. eHEALS: The eHealth Literacy Scale. J Med Internet Res. 2006 Nov 14;8(4):e27. doi: 10.2196/jmir.8.4.e27. PMID 17213046
- [Background] Porreca A, Noale M, Artibani W, Bassi PF, Bertoni F, Bracarda S, Conti GN, Corvo R, Gacci M, Graziotti P, Magrini SM, Mirone V, Montironi R, Muto G, Pecoraro S, Ricardi U, Russi E, Tubaro A, Zagonel V, Crepaldi G, Maggi S; Pros-IT CNR study group. Disease-specific and general health-related quality of life in newly diagnosed prostate cancer patients: the Pros-IT CNR study. Health Qual Life Outcomes. 2018 Jun 13;16(1):122. doi: 10.1186/s12955-018-0952-5. PMID 29898750
- [Background] Rhodes RE, Courneya KS. Investigating multiple components of attitude, subjective norm, and perceived control: an examination of the theory of planned behaviour in the exercise domain. Br J Soc Psychol. 2003 Mar;42(Pt 1):129-46. doi: 10.1348/014466603763276162. PMID 12713760
- [Background] Rhodes RE, Blanchard CM, Matheson DH. A multicomponent model of the theory of planned behaviour. Br J Health Psychol. 2006 Feb;11(Pt 1):119-37. doi: 10.1348/135910705X52633. PMID 16480559
- [Background] Trinh L, Arbour-Nicitopoulos KP, Sabiston CM, Berry SR, Loblaw A, Alibhai SMH, Jones JM, Faulkner GE. RiseTx: testing the feasibility of a web application for reducing sedentary behavior among prostate cancer survivors receiving androgen deprivation therapy. Int J Behav Nutr Phys Act. 2018 Jun 7;15(1):49. doi: 10.1186/s12966-018-0686-0. PMID 29880049
- [Background] Tudor-Locke C, Han H, Aguiar EJ, Barreira TV, Schuna JM Jr, Kang M, Rowe DA. How fast is fast enough? Walking cadence (steps/min) as a practical estimate of intensity in adults: a narrative review. Br J Sports Med. 2018 Jun;52(12):776-788. doi: 10.1136/bjsports-2017-097628. PMID 29858465
- [Background] Tudor-Locke C, Ducharme SW, Aguiar EJ, Schuna JM Jr, Barreira TV, Moore CC, Chase CJ, Gould ZR, Amalbert-Birriel MA, Mora-Gonzalez J, Chipkin SR, Staudenmayer J. Walking cadence (steps/min) and intensity in 41 to 60-year-old adults: the CADENCE-adults study. Int J Behav Nutr Phys Act. 2020 Nov 10;17(1):137. doi: 10.1186/s12966-020-01045-z. PMID 33168018
- [Background] Visser M, Koster A. Development of a questionnaire to assess sedentary time in older persons--a comparative study using accelerometry. BMC Geriatr. 2013 Jul 30;13:80. doi: 10.1186/1471-2318-13-80. PMID 23899190
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Derived] Trinh L, Sabiston CM, Alibhai SMH, Jones JM, Arbour-Nicitopoulos KP, Mina DS, Campbell K, Faulkner GE. A distance-based, randomized controlled trial for reducing sedentary behavior among prostate cancer survivors: a study protocol. BMC Public Health. 2022 Apr 28;22(1):855. doi: 10.1186/s12889-022-13218-5. PMID 35484523